CLINICAL TRIAL: NCT05752851
Title: Nanjing First Hospital，Nanjing Medical University
Brief Title: The Alteration of Gut Microbiota and Analysis of Related Factors in Newly Diagnosed Type 2 Diabetes Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20230116-10
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fecal
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T2DM group: Collect stool and blood samples，No drugs use.
- Control group: Collect stool and blood samples，No drugs use.

SUMMARY:
This Study aims to compare the characteristics of gut microbiota between the newly diagnosed T2DM and healthy subjects, and analysis the related clinical indicators that may affect the composition of gut microbiota.

DETAILED DESCRIPTION:
Previous studies have shown that gut microbiota imbalance is closely related to a variety of diseases, such as inflammatory bowel diseases (IBD), colorectal cancer (CRC), Alzheimer's disease (AD) and cardiovascular diseases. In recent years, more and more studies have found that gut microbiota plays an important role in chronic metabolic diseases such as obesity, fatty liver and diabetes. gut microbiota disorder may lead to insulin resistance，pancreatic islets injury and disorder of glycolipid metabolism through multiple metabolic pathways such as endotoxin, short chain fatty acids, bile acids, amino acids, promote the occurrence and development of T2DM. At present, there are relatively few population-based studies to assess the relationship between gut microbiota and diabetes, and the results are inconsistent or even contradictory, which may be due to the influence of the research population, disease status, diet, drugs and even detection technology. Therefore, the purpose of this study is to explore the difference of intestinal microbial characteristics between the initially diagnosed T2DM and the control group by using 16S rRNA gene sequencing analysis technology, so as to increase the understanding of the possible relationship between T2DM and intestinal microbiota, and provide theoretical support and direction guidance for the future biological treatment of diabetes.

ELIGIBILITY:
Inclusion Criteria:

1）18-65 years old 2）have no history of diabetes 3）fasting blood glucose <5.6 mmol/L 4) HbA1c<6.0%.

Exclusion Criteria:

1）BMI≥28kg/m2 2) People with type 1 diabetes, special type diabetes and pregnancy diabetes 3) Use antispasmodics, expanders, probiotics, prebiotics, antibacterial drugs or other drugs that affect intestinal microorganisms in the past month 4) Having inflammation, tumor, ulcer and other intestinal organic diseases, tumor, etc 5) History of abdominal surgery or gastrointestinal surgery 6) Suffer from mental illness or alcoholism, drug abuse or drug abuse. 7) Combined with other serious systemic diseases, such as cardiovascular disease, digestive disease, endocrine disease, skin disease, autoimmune disease, tumor, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: T2DM patients who are not treated with any hypoglycemic drugs visited in the Department of Endocrinology at the Nanjing First Hospital from January 2023 to March 2023 were enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Fecal 16S rRNA gene sequencing | Day one
  Fecal 16S rRNA gene sequencing results of two group

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Ma, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided